CLINICAL TRIAL: NCT02006576
Title: Proof-of-concept Study to Demonstrate Inhibition of Prostaglandin E (PGE) Production and Associated Biological Effects in the Lower Respiratory Tract by Ibuprofen.
Brief Title: Prostaglandin Inhibition for Emphysema
Acronym: PIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Jewish Health (Other); Temple University (Other); University of California, Los Angeles (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0503-13-ET
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Emphysema
Keywords: Emphysema; Prostaglandin E; Bronchoalveolar lavage
MeSH Terms: conditions — Emphysema | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- COPD, Placebo (Placebo Comparator): Placebo three times daily
  Interventions: Other: Placebo three times daily
- Control subject (No Intervention): Control subjects, no intervention
- COPD, ibuprofen (Experimental): 600 mg ibuprofen three times daily for 48 weeks
  Interventions: Drug: 600 mg ibuprofen three times daily for 48 weeks

INTERVENTIONS:
Drug: 600 mg ibuprofen three times daily for 48 weeks
  Other Names: Advil, Children's Ibuprofen, Advil Migraine, Motrin IB, NeoProfen, Caldolor, Wal-Profen, I-Prin
  Arms: COPD, ibuprofen
Other: Placebo three times daily
  Arms: COPD, Placebo

SUMMARY:
The Prostaglandin Inhibition for Emphysema (PIE) study will determine if a currently available therapy, ibuprofen 600 mg three times daily, can block PGE production in the lower respiratory tract and if this results in improvement in measures of lung repair function.

DETAILED DESCRIPTION:
The Prostaglandin Inhibition for Emphysema (PIE) study will determine if a currently available therapy, ibuprofen 600 mg three times daily, can block PGE production in the lower respiratory tract and if this results in improvement in measures of lung repair function. This is a proof-of-concept study. The PIE study will set the stage for novel therapy to modify the course of chronic obstructive pulmonary disease (COPD).

COPD is the third leading cause of death in the United States. No currently available treatment can meaningfully restore lung function that is lost in this disease. Emphysema is a major component of COPD and results when lung damage exceeds the ability of the lung to repair. Recent evidence indicates that the repair processes present in the normal lung are deficient in patients with emphysema and that this is due, in part, to suppression of repair by an inflammatory mediator: prostaglandin E (PGE). Currently available therapies can block PGE production, but whether this can be achieved in the lung in COPD is unknown. The PIE study will answer that question.

This will be accomplished by performing a randomized, double blind, placebo-controlled, parallel group study that will compare a widely used and well-tolerated non-steroidal anti-inflammatory drug, ibuprofen 600 mg three times daily, with placebo. PGE will be measured directly in the lower respiratory tract by sampling the lung with the technique of bronchoalveolar lavage. Secondary measures will be made, quantifying PGE in induced sputum and quantifying PGE metabolites in blood and urine. In addition, the current proposal will determine if biochemical measures of lung repair are restored by treatments that block PGE production. Additional outcomes will also be assessed including the effect of treatment on PGD and other eicosanoids and assessing IL-8 and neutrophils in sputum and BAL fluid and selected inflammatory biomarkers present in serum that may be associated with lung function decline. Finally, in an accompanying Ancillary Study, the current proposal will determine if alveolar macrophages over-produce PGE and/or PGD in COPD and will determine if the microRNA miR-146a modulates the production of these prostaglandins, as we have demonstrated for lung fibroblasts. The Ancillary Study will also determine if genetic variation in a miR-146a is related to differential expression.

The proposed research will, therefore, determine if inhibition of PGE production can be achieved in the lung, if this appears to restore lung repair mechanisms and will help determine who would benefit from such a therapeutic approach. This is a highly novel approach to the treatment of emphysema and has the potential to restore lost lung function, a crucial unmet medical need for a major public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Age > 45 years
* Emphysema (>5% of voxels <950 Hounsfield Units determined on the CT scan performed as part of the COPDGene study as quantified at the COPDGene radiology center). An equivalent scan as determined by the radiology center is also acceptable.
* Post-bronchodilator FEV1 > 35% predicted)
* Smoker or ex-smoker (10 pack years minimum)

Exclusion Criteria:

* Contraindication to bronchoscopy or other study procedures
* Pregnancy of plans to become pregnant within six months
* Aspirin-sensitive asthma
* Regular use of systemic glucocorticoid
* Regular use of an NSAID (low dose aspirin for cardiac disease is acceptable and subjects taking only this regularly will be eligible)
* Unstable medical condition
* History of myocardial infarction or unstable angina within six months
* Allergy to or history of adverse effect from ibuprofen or other NSAID
* History of gastrointestinal bleeding within one year
* Any condition that, in the opinion of the investigator, places the subject at untoward risk
* Inability to provide informed consent

Ages: 46 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I Rennard, MD, Study Chair — University of Nebraska
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harbor-UCLA Medical Center, Torrance, California
  - National Jewish Health, Denver, Colorado
  - Univerisity of Nebraska Medical Center, Omaha, Nebraska
  - Temple University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COPD, Placebo | Control Subject | COPD, Ibuprofen
Started | 35 | 51 | 32
Completed | 17 | 44 | 15
Not Completed | 18 | 7 | 17
Not completed — Withdrawal by Subject | 4 | 6 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Screen Failure, too sick, other | 13 | 1 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COPD, Placebo | Control Subject | COPD, Ibuprofen | Total
Number analyzed (Participants) | 35 | 51 | 32 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 37 | 17 | 75
  >=65 years | 14 | 14 | 15 | 43
Age, Continuous [Median (Full Range); unit: years] | 63.8 [49.3 to 81.9] | 58.8 [50.0 to 78.5] | 63.9 [52.9 to 78.0] | 60.9 [49.3 to 81.9]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex is missing for one person.
  Participants
    number analyzed (Participants) | 35 | 51 | 31 | 117
    Female | 16 | 24 | 15 | 55
    Male | 19 | 27 | 16 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 21 | 9 | 41
  White | 12 | 27 | 11 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 3 | 12 | 27
Region of Enrollment [Number; unit: participants]
  United States | 35 | 51 | 32 | 118

OUTCOME MEASURES:

1. Primary Outcome: Will Ibuprofen, 600 mg Three Times Daily, Decrease PGE Concentration in the Alveolar Portion of BAL Fluid in Subjects With Emphysema in Comparison to Placebo?
Description: PGE will be measured by HPLC in alveolar fluids obtained at randomization (week 0) and again 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group.
Time Frame: 12 weeks after subject randomization
Population: Primary analysis limited to COPD Placebo vs. Ibuprofen groups only. The 'control' group is assessed once and serves as a comparator for the post treatment ibuprofen group.
Measure: Mean (Standard Deviation); unit: Change in ng/ml
Arm/Group | COPD, Placebo | Control Subject | COPD, Ibuprofen
Number analyzed (Participants) | 17 | 0 | 15
Change in ng/ml | 0.003 (0.080) |  | -0.156 (0.455)

2. Secondary Outcome: Will Ibuprofen, 600 mg Three Times Daily, Increase Pro-collagen Peptide Fragment Concentrations in the Alveolar Portion of BAL Fluid in Subjects With Emphysema in Comparison to Placebo?
Description: Pro-collagen peptide fragments will be measured by ELISA in alveolar fluids obtained at randomization (week 0) and again 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group.
Time Frame: 12 weeks after subject randomization
Population: This analysis limited to COPD Placebo vs. Ibuprofen groups only.
Measure: Mean (Standard Deviation); unit: Change in ng/ml
Arm/Group | COPD, Placebo | Control Subject | COPD, Ibuprofen
Number analyzed (Participants) | 16 | 0 | 13
Change in ng/ml | -1.060 (8.729) |  | 0.011 (0.584)

3. Other Pre Specified Outcome: Prostaglandin E Concentrations n Participants With Emphysema v in Smoking, Former Smoking and Healthy Non-smoking Controls After Ibuprofen Three Times Daily
Description: Comparing ibuprofen, 600 mg three times daily, in reducing prostaglandin E concentrations in the alveolar portion of bronchoalveolar lavage (BAL) fluid in participants with emphysema to those present in smoking, former smoking and healthy non-smoking controls? Prostaglandin E (PGE) will be measured by HPLC in alveolar fluids obtained at randomization and again 12 weeks after randomization on subjects taking ibuprofen to compare emphysema subjects, smokers, former smokers and controls.
Time Frame: 12 weeks after subject randomization
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce Prostaglandin E Concentrations in the Bronchial Portion of BAL Fluid in Subjects With Emphysema Compared to Placebo?
Description: PGE will be measured by HPLC in bronchial fluids obtained at randomization and again 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after subject randomization
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce Prostaglandin E Concentrations in Induced Sputum From Subjects With Emphysema Compared to Placebo?
Description: PGE will be measured by HPLC in sputum samples obtained prior to randomization and again 10 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smokers and controls.
Time Frame: 10 weeks after subject randomization
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce the PGE Metabolite PGEM in the Peripheral Blood of Subjects With Emphysema Compared to Placebo?
Description: PGEM will be measured by HPLC in peripheral blood specimens obtained at randomization, 12 weeks after randomization and 48 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce the PGE Metabolite PGEM in the Urine of Subjects With Emphysema Compared to Placebo?
Description: PGEM will be measured by HPLC in urine specimens obtained at randomization, 12 weeks after randomization and 48 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Will Ibuprofen, 600 mg Three Times Daily, Increase Pro-collagen Peptide Fragment Concentrations in the Alveolar Portion of BAL Fluid in Subjects to the Range Observed in Normal Individuals or to Higher Levels?
Description: Pro-collagen peptide fragment concentrations will be measured by ELISA in alveolar fluids obtained at randomization and again 12 weeks after randomization to determine if levels reach those of normal individuals or reach even higher levels.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Increase the Procollagen III Amino Peptide Excreted Into the Urine of Subjects With Emphysema Compared to Placebo?
Description: Procollagen III amino peptide will be measured by ELISA in urine specimens obtained at randomization, 12 weeks after randomization and 48 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Will Ibuprofen, 600 mg Three Times Daily, Decrease IL-8 Concentrations in the Alveolar Portion of BAL Fluid in Subjects With Emphysema in Comparison to Placebo?
Description: IL-8 will be measured by ELISA in alveolar specimens obtained at randomization and 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Will Ibuprofen, 600 mg Three Times Daily, Decrease Neutrophil Concentrations in the Alveolar Portion of BAL Fluid in Subjects With Emphysema in Comparison to Placebo?
Description: Neutrophils will be measured by 500 cell differentials in alveolar specimens obtained at randomization and 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce IL-8 Concentrations in the Bronchial Portion of BAL Fluid in Subjects With Emphysema Compared to Placebo?
Description: IL-8 will be measured by ELISA in bronchial specimens obtained at randomization and 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce IL-8 Concentrations in Induced Sputum From Subjects With Emphysema Compared to Placebo?
Description: IL-8 will be measured by ELISA in sputum specimens obtained prior to randomization and 10 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 10 weeks after randomization
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce PMN Concentrations in the Bronchial Portion of BAL Fluid in Subjects With Emphysema Compared to Placebo?
Description: Neutrophils will be measured by 500 cell differentials in bronchial specimens obtained at randomization and 12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce PMN Concentrations in Induced Sputum From Subjects With Emphysema Compared to Placebo?
Description: Neutrophils will be measured by 500 cell differentials in bronchial specimens obtained prior to randomization and 10 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 10 weeks after randomization
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Alter LTB4 Concentrations in Subjects With Emphysema Compared to Placebo in the Alveolar Portion of BAL, Bronchial Portion of BAL and Induced Sputum?
Description: LTB4 will be measured by HPLC in alveolar fluids, bronchial fluids and induced sputums obtained at randomization and again 10-12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce Concentrations of CC-16 in Serum From Subjects With Emphysema Compared to Placebo?
Description: CC-16 will be measured by ELISA in serum specimens obtained at randomization, 12 weeks after randomization and 48 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce Concentrations of CRP in Serum From Subjects With Emphysema Compared to Placebo?
Description: CRP will be measured by ELISA in serum specimens obtained at randomization, 12 weeks after randomization and 48 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce Concentrations of SP-d in Serum From Subjects With Emphysema Compared to Placebo?
Description: SP-d will be measured by ELISA in serum specimens obtained at randomization, 12 weeks after randomization and 48 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Are Levels of PGD Increased in the Alveolar Component of BAL Fluid in Patients With COPD? Are Levels of PGD in Alveolar Lavage Fluid Related to FEV1 and/or Severity of Emphysema?
Description: PGD will be measured by HPLC in alveolar fluids obtained at randomization and again 10-12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls. PGD levels will be compared against FEV1 and severity of emphysema.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Are Levels of TXB2 (the Primary Metabolite of Thromboxane) Increased in the Alveolar Component of BAL Fluid in Patients With COPD? Are the Levels Related to FEV1 and/or Severity of Emphysema?
Description: TXB2 will be measured by HPLC in alveolar fluids obtained at randomization and again 10-12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls. TXB2 levels will be compared against FEV1 and severity of emphysema.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Are Levels of 6kPGF1a (the Primary Metabolite of Prostacyclin) Increased in the Alveolar Component of BAL Fluid in Patients With COPD? Are the Levels Related to FEV1 and/or Severity of Emphysema?
Description: 6kPGF1a will be measured by HPLC in alveolar fluids obtained at randomization and again 10-12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls. 6kPGF1a levels will be compared against FEV1 and severity of emphysema.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily, Reduce the Eicosanoids Other Than PGE in Subjects With Emphysema Compared to Placebo in BAL and Induced Sputum?
Description: LTB4, PGD, TXB2, and 6kPGF1a will be measured by HPLC in induced sputums and BAL's obtained prior to randomization and again 10-12 weeks after randomization on emphysema subjects taking placebo and emphysema subjects taking ibuprofen to compare control group versus treatment group. The emphysema group will also be compared to smokers, former smoker, and controls.
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily Alter the Rate of Change of Emphysema Progression as Assessed by CT Scan?
Description: CT scans will be used to evaluated the rate of change of emphysema for participants taking 600 mg of ibuprofen three times a day
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily Alter the Rate of Change of DLCO?
Description: Spirometry will be used to test lung function [diffusing capacity of the lungs for carbon monoxide (DLCO)] to assess the lungs' ability to transfer gas from inspired air to the bloodstream in participants taking 600 mg of ibuprofen three times a day.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily Alter the Rate of Change of FEV1?
Description: Evaluation of 600 mg of Ibuprofen three times a day on forced expiratory volume (FEV1) rate of change. FEV1 calculates the amount of air that a person can force out of their lungs in 1 second. FEV1 values that are lower than average suggest the presence of COPD.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily Alter the Rate of COPD Exacerbations?
Description: Evaluation of the rate of chronic obstructive pulmonary disease (COPD) exacerbations in participants taking 600 mg of Ibuprofen three times a day.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Will Ibuprofen 600 mg Three Times Daily Alter Health Status Assessed by the SGRQ or COPD Status Assessed by the CAT in Participants With Emphysema ?
Description: Evaluation of 600 mg of Ibuprofen three times a day on health status of participants with emphysema as assessed by St. George's Respiratory Questionnaire (SGRQ) or chronic obstructive pulmonary disease (COPD) status as assessed by computed axial tomography (CAT). St. George's Respiratory Questionnaire (SGRQ) is a type of questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Chronic obstructive pulmonary disease, or COPD, refers to a group of diseases that cause airflow blockage and breathing-related problems. It includes emphysema and chronic bronchitis.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Are There Differences Between Subjects With Upper Lobe vs. Lower Lobe Emphysema?
Description: PGE levels in BAL fluid, sputum and metabolites in blood and urine will be evaluated for differences between subjects with upper lobe vs. lower lobe emphysema. Procollagen peptides will be evaluated in BAL fluid between subjects with upper lobe vs. lower lobe emphysema. Eicosanoids (PGD, 6kPGF1a, TXB2) urine will be evaluated between subjects with upper lobe vs. lower lobe emphysema. Measures of inflammation will be evaluated between subjects with upper vs. lower lobe emphysema. Does the response of PGE, measures of repair, response of other eicosanoids, and response of measures of inflammation change as a result of 600 mg three times daily of ibuprofen.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Are There Differences Between Subjects With Clustered vs. Diffuse Emphysema?
Description: PGE levels in BAL fluid, sputum and metabolites in blood and urine will be evaluated for differences between subjects with clustered versus diffuse emphysema. Procollagen peptides will be evaluated in BAL fluid between subjects with clustered versus diffuse emphysema. Eicosanoids (PGD, 6kPGF1a, TXB2) urine will be evaluated between subjects with clustered versus diffuse emphysema. Measures of inflammation will be evaluated between subjects with clustered versus diffuse emphysema. Does the response of PGE, measures of repair, response of other eicosanoids, and response of measures of inflammation change as a result of 600 mg three times daily of ibuprofen.
Time Frame: 48 weeks after randomization
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Will BAL PGE Levels be Related to the Rate of Emphysema Progression Determined by the Change in Computed Tomography (CT) Quantified Lung Density in COPDGene?
Description: Evaluation of prostaglandin E (PGE) levels obtained by bronchoalveolar lavage (BAL) and emphysema progression as determined by change in computed tomography (CT) quantified lung density.
Time Frame: 3-6 years from initial CT scan
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Will BAL PGE Levels Assessed at Study Initiation be Related to the Rate of Emphysema Progression Determined by the Change in FEV1 From the Time of Assessment in COPDGene?
Description: Evaluation of prostaglandin E (PGE) levels obtained by bronchoalveolar lavage (BAL) and emphysema progression as determined by change in forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. FEV1 values that are lower than average suggest the presence of COPD.
Time Frame: 3-6 years from initial FEV1 assessment
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Will Measures of Prostanoids be Related to the Rate of Emphysema Progression Determined by the Change in CT Quantified Lung Density in COPDGene?
Description: Comparing measures of prostanoids, other than PGE, to the rate of emphysema progression as determined by the change in computed tomography (CT) quantified lung density from assessment to end of study.
Time Frame: 3-6 years from initial CT scan
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Will Measures of Inflammation Assessed at Study Initiation be Related to the Rate of Emphysema Progression Determined by the Change in FEV1 From the Time of Assessment in COPDGene
Description: Emphysema progression as determined by the change in forced expiratory volume (FEV1) from assessment to end of study. FEV1 calculates the amount of air that a person can force out of their lungs in 1 second. FEV1 values that are lower than average suggest the presence of COPD.
Time Frame: 3-6 years after initial FEV1 assessment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Three year period from the first study visit through the last completed study visit on at 48 weeks.
Arm/Group | COPD, Placebo | Control Subject | COPD, Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/51 | 1/32
Serious Adverse Events (participants affected / at risk) | 4/35 | 0/51 | 2/32
Other Adverse Events (participants affected / at risk) | 4/35 | 0/51 | 11/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPD, Placebo (N=35) | Control Subject (N=51) | COPD, Ibuprofen (N=32)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Left Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPD, Placebo (N=35) | Control Subject (N=51) | COPD, Ibuprofen (N=32)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Headache (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Positive Occult Blood (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
AECOPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Acute Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mild benign-appearing intrinsic stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Left Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Viral Gastroenteresis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough and Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02006576/Prot_SAP_000.pdf